CLINICAL TRIAL: NCT03299179
Title: The Effects of the Female Sex Hormones and Hormonal Contraception on Cerebral Perfusion
Brief Title: The Effects of the Female Hormones on Cerebral Perfusion
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2016/0757
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Perfusion; Contraception; Menstrual Cycle
MeSH Terms: interventions — Magnetic Resonance Imaging; Monitoring, Physiologic; Blood Specimen Collection; Blood Pressure Determination; Body Temperature; Surveys and Questionnaires; Pregnancy Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural cycle: 15 female volunteers, not using hormonal contraception, will be scanned during 3 menstrual cycles. During each cycle, the volunteers will be scanned 3 times: during the follicular phase, during ovulation and during luteal phase.
  Interventions: Device: MRI scan; Device: Physiological monitoring; Biological: Blood sample; Device: Blood pressure measurement; Device: Body temperature; Other: Questionnaires; Diagnostic Test: Pregnancy test
- Anti-conception: 15 female volunteers, using hormonal contraception pill Deso 20, will be scanned during 3 menstrual cycles. During each cycle, the volunteers will be scanned 2 times: during the pill-week and during the pill-free week.
  Interventions: Device: MRI scan; Device: Physiological monitoring; Biological: Blood sample; Device: Blood pressure measurement; Device: Body temperature; Other: Questionnaires

INTERVENTIONS:
Device: MRI scan — Several MRI scan modalities: MPRAGE (structural scan), arterial spin labeling (cerebral perfusion), resting state functional-MRI (fMRI, cerebral activity) and diffusion MRI (white matter diffusion and white matter tracts).
Device: Physiological monitoring — During MRI: heart rate, end-tidal carbon dioxide (CO2), respiratory rate and skin conductance
Biological: Blood sample — Blood sample after MRI-session: measurement of hematocrit, hemoglobin, estradiol, progesterone, follicle stimulation hormone and luteinizing hormone.
Device: Blood pressure measurement — Measuring blood pressure before and after MRI-scan
Device: Body temperature — Measuring body temperature before and after MRI-scan
Other: Questionnaires — Questionnaires at the start of the study on lifestyle. Additionally, a questionnaire before each scan session on the actual state of the volunteer (e.g. mood, caffeine consumption, alcohol, medication, etc.)
Diagnostic Test: Pregnancy test — Test for pregnancy using a pregnancy dipstick test
  Groups: Natural cycle

SUMMARY:
Measuring brain perfusion is biased by a inter- and intrasubject variability, caused by physiological and lifestyle factors. In this study, the investigators want to investigate the variations in cerebral perfusion and other brain parameters (grey matter, resting-state brain activity, brain connectivity and white matter diffusion) caused by the female sex hormones and hormonal contraception.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor or Master student
* Minimum of 3 months not using contraception of using Deso20

Exclusion Criteria:

* No informed consent
* MRI-contraindications
* Claustrophobia
* Pregnancy or breastfeeding
* Chronic diseases and chronic medication use
* Smoker
* Drug use
* Abuse of alcohol and caffeine

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 healthy young volunteers, either using no hormonal anti-conception, either using Deso20 as anti-conception.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2016-10-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional cerebral perfusion (ml/100g/min): natural versus contraception | measured during scan-session
  Differences in regional perfusion between volunteers of the natural cycle group versus the volunteers using contraception
Regional cerebral perfusion (ml/100g/min) variations during natural menstrual cycle | measured during scan-session
  Variations in cerebral perfusion during the menstrual cycle: follicular phase versus ovulation versus luteal phase in the natural cycle group, correlated with female hormones measured in blood sample
Regional cerebral perfusion (ml/100g/min) variations during menstrual cycle using contraception | measured during scan-session
  Variations in cerebral perfusion during the menstrual cycle: pill-week versus pill-free week in the contraception group, correlated with female hormones measured in blood sample

SECONDARY OUTCOMES:
Regional grey matter volume (mm³): natural versus contraception | measured during scan-session
  Differences in regional grey matter volume between volunteers of the natural cycle group versus the volunteers using contraception
Regional grey matter volume (mm³) variations during natural menstrual cycle | measured during scan-session
  Variations during the menstrual cycle: follicular phase versus ovulation versus luteal phase in the natural cycle group, correlated with female hormones measured in blood sample
Regional grey matter volume (mm³) variations during menstrual cycle using contraception | measured during scan-session
  Variations in grey matter volume during the menstrual cycle: pill-week versus pill-free week in the contraception group, correlated with female hormones measured in blood sample
Resting state brain activity: natural versus contraception | measured during scan-session
  Differences in resting state brain activity between volunteers of the natural cycle group versus the volunteers using contraception
Resting state brain activity variations during natural menstrual cycle | measured during scan-session
  Variations in resting state brain activity during the menstrual cycle: follicular phase versus ovulation versus luteal phase in the natural cycle group, correlated with female hormones measured in blood sample
Resting state brain activity variations during menstrual cycle using contraception | measured during scan-session
  Variations in resting state brain activity during the menstrual cycle: pill-week versus pill-free week in the contraception group, correlated with female hormones measured in blood sample
Cerebral diffusion properties: natural versus contraception | measured during scan-session
  Differences in diffusion properties (Mean Diffusivity(MD)/Apparent Diffusion Coefficient (ADC)/fractional Anisotropy(FA)) between volunteers of the natural cycle group versus the volunteers using contraception
Cerebral diffusion properties variations during natural menstrual cycle | measured during scan-session
  Variations in diffusion properties (MD/ADC/FA) during the menstrual cycle: follicular phase versus ovulation versus luteal phase in the natural cycle group, correlated with female hormones measured in blood sample
Cerebral diffusion properties variations during menstrual cycle using contraception | measured during scan-session
  Variations in diffusion properties (MD/ADC/FA) during the menstrual cycle: pill-week versus pill-free week in the contraception group, correlated with female hormones measured in blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Eric Achten, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided